CLINICAL TRIAL: NCT03751683
Title: Evaluation Genotypic, Phenotypic and Prognosis Autoimmune Polyendocrinopathy Candidiasis Ectodermal Dystrophy (APECED) Syndrome
Brief Title: Evaluation Genotypic, Phenotypic and Prognosis APECED Syndrome
Acronym: APECED
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2008_30/0915; 2009-A00197-50 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2018-11-21; First posted 2018-11-23 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: APECED
MeSH Terms: conditions — Polyendocrinopathies, Autoimmune

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of the study will define the mutational spectrum in this French cohort, in patients with APECED syndrome genetically authenticated

ELIGIBILITY:
Inclusion Criteria:

* patients with at least 2 major criteria out of the following 3: hypoparathyroidism of autoimmune origin, adrenal insufficiency of autoimmune origin, chronic cutaneous and mucosal candidiasis.
* patients with only 1 of the 3 major criteria, associated with at least 2 of the following minor criteria: hypergonadotropic hypogonadism of autoimmune origin, atrophic gastritis, malabsorption, autoimmune hepatitis, vitiligo, alopecia, chronic keratoconjunctivitis, hypoplasia of dental enamel.
* patients whose molecular diagnosis has been established or who will be established during the inclusion visit with the genetic sample.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A patient diagnosed or suspected of a genetic disorder of immunity control, known as APECED syndrome (Autoimmune Polyendocrinopathy Candidiasis Ectodermal Dystrophy) or autoimmune polyendocrinopathy type 1,
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2009-07-30 (Actual); Primary Completion 2018-01-25 (Actual); Study Completion 2018-01-25 (Actual)

PRIMARY OUTCOMES:
allelic frequency of the mutation c.967-979del13 of the AIRE gene | Baseline: one session

SECONDARY OUTCOMES:
total number of cases recognized APECED syndrome regardless of the diagnostic criteria used. | Baseline: one session
correlations between the clinical phenotype and the autoantibodies on all cases with APECED syndrome. | Baseline: one session
correlations between the mutations of the AIRE gene and the HLA genotyping on all cases with APECED syndrome. | Baseline: one session
prevalence of types of antibodies found on APECED syndrome. | Baseline: one session
the distribution of lymphocyte subpopulations on the whole cases with APECED syndrome. | Baseline: one session
proportion of patients with a molecular diagnosis of positive APECED syndrome, among patients presenting our new diagnostic criteria (a major criterion and at least 2 criteria | Baseline: one session

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuelle Proust-Lemoine, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- CHRU, Hôpital Claude Huriez, Lille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Humbert L, Proust-Lemoine E, Dubucquoi S, Kemp EH, Saugier-Veber P, Fabien N, Raymond-Top I, Cardot-Bauters C, Carel JC, Cartigny M, Chabre O, Chanson P, Delemer B, Do Cao C, Guignat L, Kahn JE, Kerlan V, Lefebvre H, Linglart A, Mallone R, Reynaud R, Sendid B, Souchon PF, Touraine P, Wemeau JL, Vantyghem MC. Lessons From Prospective Longitudinal Follow-up of a French APECED Cohort. J Clin Endocrinol Metab. 2025 Feb 18;110(3):e757-e773. doi: 10.1210/clinem/dgae211. PMID 38605470